CLINICAL TRIAL: NCT05244681
Title: Experiences of a Home-based Virtual Reality Serious Game in People With Chronic Non-specific Neck Pain: A Qualitative Study.
Brief Title: Experiences of a Home-based Virtual Reality Serious Game in People With Chronic Non-specific Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Collaborators: Fonds National de la Recherche Scientifique (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: VR NECK PAIN
Record Dates: First submitted 2022-02-07; First posted 2022-02-17 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Chronic Non-specific Neck Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- People with chronic non-specific neck pain (Other): Group of people with chronic non-specific neck pain who agreed to participate in a semi-structured interview about their experience using an immersive virtual reality serious game at home
  Interventions: Other: Semi-structured interview

INTERVENTIONS:
Other: Semi-structured interview — Semi-structured interview to explore the experience of people with chronic non-specific neck pain who used an immersive virtual reality serious game at home

SUMMARY:
Background: Immersive virtual reality (VR) has been used for several years in the treatment of chronic neck pain. This new type of rehabilitation device, which can be used at home, is promising and seems to be as effective as conventional treatments for neck pain. Exploring the experience of people with chronic neck pain using this type of rehabilitation device at home could, among other things, help to understand the factors favoring good adherence and those not favoring it. This could also help us to improve VR home rehabilitation programs according to the patients' needs, preferences and expectations. However, currently, no studies have qualitatively evaluated the experience of people with chronic non-specific neck pain using an immersive VR serious game at home.

Objective: To explore the experience of people with chronic non-specific neck pain who used an immersive VR serious game at home.

Methods: Individual semi-structured interviews will be conducted with people with chronic non-specific neck pain. Interviews will last for approximately 30 to 60 minutes and will be carried out face-to-face or via videoconference (Microsoft Teams), depending on up-to-date guidance relating to the Covid-19 pandemic. Semi-structured interviews will be audio-recorded and transcribed verbatim. The transcripts will be read several times and analyzed using thematic analysis, with themes emerging from the transcripts (inductive approach). These themes will be defined and revised throughout the analysis process.

Discussion: Study findings will help to better understand the experience of people with chronic non-specific neck pain using a VR serious game at home, and then will allow to adapt it to the subjects' needs, preferences and expectations. These adaptations could further increase adherence to treatment and/or improve clinical outcomes for people with chronic non-specific neck pain using this type of rehabilitation device at home.

ELIGIBILITY:
Inclusion Criteria:

* Adults (over 18 years), men or women, living in Belgium
* Chronic (> 3 months) non-specific neck pain (no specific cause responsible for the neck pain)
* To speak fluent French and to be able to provide informed consent to take part in an interview
* To be able to take part in a semi-structured interview
* No susceptibility to motion sickness, according to the Motion Sickness Susceptibility Questionnaire (MSSQ)

Exclusion Criteria:

* Age under 18 years
* Specific cause responsible for the neck pain (cancer, fracture, etc.)
* Signs of sensorimotor dysfunction (dizziness, vestibular disorders)
* Susceptibility to motion sickness, according to the MSSQ
* Vision problems
* Altered comprehension or inability to speak fluent French
* Inability to provide written informed consent or to take part in a semi-structured interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
General experience with the virtual reality serious game | 30-60 minutes
  Participants' responses based on the questions asked in the semi-structured interviews

CONTACTS AND LOCATIONS:
Overall Officials: Christine Detrembleur, PhD, Principal Investigator — Université Catholique de Louvain
Locations (1):
- Université Catholique de Louvain, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No